CLINICAL TRIAL: NCT01938625
Title: Phase 2, Open-Label Study to Investigate the Pharmacokinetics, Efficacy, Safety, and Tolerability of the Combination of Simeprevir (TMC435), Daclatasvir (BMS-790052) and Ribavirin (RBV) in Subjects With Recurrent Chronic Hepatitis C Genotype 1b Infection After Orthotopic Liver Transplantation
Brief Title: A Study of Pharmacokinetics, Efficacy, Safety, Tolerability, of the Combination of Simeprevir (TMC435), Daclatasvir (BMS-790052), and Ribavirin (RBV) in Patients With Recurrent Chronic Hepatitis C Genotype 1b Infection After Orthotopic Liver Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR102639; TMC435HPC3016 (Other: Janssen R&D Ireland); 2013-002726-23 (EudraCT Number)
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; Recurrent Chronic Hepatitis C; Pharmacokinetics; Simeprevir; Daclatasvir; Ribavirin; Orthotopic Liver Transplantation; TMC435; BMS-790052; RBV
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Simeprevir; daclatasvir; Ribavirin; Cyclosporine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): Participants with Metavir fibrosis score F1-F2 will receive treatment with combinational regimen of simeprevir, daclatasvir, and ribavirin along with cyclosporine or tacrolimus as stable immunosuppressant therapy.
  Interventions: Drug: Simeprevir; Drug: Daclatasvir; Drug: Ribavirin; Drug: Cyclosporine; Drug: Tacrolimus
- Part 2 (Experimental): Participants with Metavir fibrosis score F1-F4 will receive treatment with combinational regimen of simeprevir, daclatasvir, and ribavirin along with tacrolimus as stable immunosuppressant therapy.
  Interventions: Drug: Simeprevir; Drug: Daclatasvir; Drug: Ribavirin; Drug: Tacrolimus

INTERVENTIONS:
Drug: Simeprevir — Participants will receive 150 milligram capsule of simeprevir orally (by mouth) once daily with food for 24 weeks. In Part 1, if simeprevir pre-dose plasma concentration is greater than 7,300 nanogram per milliliter (ng/mL), participants will receive simeprevir 150 milligram capsule orally every other day to complete 24 weeks of treatment.
Drug: Daclatasvir — Participants will receive 60 milligram tablet of daclatasvir orally once daily for 24 weeks.
Drug: Ribavirin — Participants will receive 5 or 6 tablets of 200 milligram of ribavirin orally twice a day with food for 24 weeks.
Drug: Cyclosporine — Participants will receive cyclosporine as one of the stable immunosuppressant therapy (no change in dose in the last month) for more than 3 months prior to the screening visit. Cyclosporine will be administered as per the manufacturer's prescribing information for 24 weeks.
  Arms: Part 1
Drug: Tacrolimus — Participants will receive tacrolimus as one of the stable immunosuppressant therapy (no change in dose in the last month) for more than 3 months prior to the screening visit. Tacrolimus will be administered as per the manufacturer's prescribing information for 24 weeks.

SUMMARY:
The purpose of the study is to evaluate effect of steady-state (when the amount of drug administered (in a given time period is equal to the amount of drug eliminated in that same period) of simeprevir and daclatasvir on the steady-state pharmacokinetics (what a medication does to the body) of cyclosporine (applicable to Part 1 only) and tacrolimus when administered as a combinational regimen in post-orthotopic liver transplantation (OLT) participants with recurrent hepatitis C virus (HCV) genotype 1b infection and effectiveness of a 24-week treatment regimen containing simeprevir, daclatasvir, and ribavirin (RBV) with respect to the proportion of HCV genotype 1b infected post-OLT participants achieving sustained virologic response 12 weeks after end of treatment.

DETAILED DESCRIPTION:
This is an open-label (all participants of this study know the identity of the intervention) and multicenter (study conducted at multiple sites) study. This study will be conducted in 2 parts. Both the parts of the study will consist of screening phase (4 weeks), treatment period (24 weeks), and a post-treatment follow-up (24 weeks). A total of 30 participants will be enrolled in Part 1 and Part 2 of the study. A minimum of 9 participants were planned to receive cyclosporine as stable immunosuppressant therapy and a minimum of 9 participants were planned to receive tacrolimus as stable immunosuppressant therapy during Part 1. All participants will be receiving tacrolimus as stable immunosuppressant therapy during Part 2. In Part 1 of the study, participants with Metavir score of F1-F2, will receive a combination of study drugs - simeprevir, daclatasvir, and ribavirin for 24 weeks. In Part 2 of the study, participants with Metavir score F1-F4 will receive a dosing regimen of study drugs based on the data from Part 1 of the study. Safety evaluations will include assessments of adverse events, clinical laboratory tests, urinalysis, electrocardiogram, vital signs, and physical examination. The total study duration for each participant will be approximately 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant between 6 months and 10 years prior to the screening visit
* Hepatitis C virus (HCV) genotype 1 subtype b infection confirmed at screening
* Screening HCV ribonucleic acid level greater than 10,000 IU/mL
* HCV treatment-naïve participants must not have received post orthotopic liver transplant treatment with any approved or investigational drug for the treatment of HCV
* Receiving stable immunosuppressant therapy (ie, no change in dose in the last month) with cyclosporine (only allowed in Part 1) or tacrolimus for more than 3 months prior to the screening visit

Exclusion Criteria:

* Evidence of acute or chronic hepatic decompensation after the liver transplantation (including ascites, bleeding varices or hepatic encephalopathy)
* Any liver disease of non-HCV etiology, including current evidence of graft rejection except the presence of liver steatosis
* Any other clinically significant disease that in the opinion of the investigator would be exacerbated by the known effects of ribavirin
* Coinfection with HCV of another genotype than genotype 1b, HIV type 1 or 2 (positive HIV-1 or HIV-2 antibodies test at screening), and hepatitis B virus (hepatitis B surface antigen positive)
* Multi-organ transplant that included heart, lung, pancreas, or kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-12-12 (Actual); Primary Completion 2015-04-27 (Actual); Study Completion 2015-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (6):
- Germany (2):
  - Essen
  - Hamburg
- Warsaw, Poland
- Spain (3):
  - Barcelona
  - Madrid
  - Valencia

REFERENCES:
- [Derived] Forns X, Berenguer M, Herzer K, Sterneck M, Donato MF, Andreone P, Fagiuoli S, Cieciura T, Durlik M, Calleja JL, Marino Z, Shukla U, Verbinnen T, Lenz O, Ouwerkerk-Mahadevan S, Peeters M, Janssen K, Kalmeijer R, Jessner W. Efficacy, safety, and pharmacokinetics of simeprevir, daclatasvir, and ribavirin in patients with recurrent hepatitis C virus genotype 1b infection after orthotopic liver transplantation: The Phase II SATURN study. Transpl Infect Dis. 2017 Jun;19(3). doi: 10.1111/tid.12696. Epub 2017 May 4. PMID 28295849

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in 2 parts (part 1 and part 2) to sequentially enroll the participants. All analyses were conducted on the overall study population (part 1 and part 2 combined).
Groups:
- Cyclosporine: Participants received simeprevir (SMV) 150 milligram (mg) once daily (qd) or once every other day (qod) as applicable with food and daclatasvir (DCV) 60 mg qd with food and ribavirin (RBV) 1000 or 1200 milligram per day (mg/day) twice daily (bid) with food for 24 Weeks along with cyclosporine as immunosuppressant therapy for more than 3 months prior to the screening visit.
- Tacrolimus: Participants received SMV 150 mg qd or qod as applicable with food and DCV 60 mg qd with food and RBV 1000 or 1200 mg/day bid with food for 24 Weeks along with tacrolimus as immunosuppressant therapy for more than 3 months prior to the screening visit.
Period: Overall Study
Arm/Group | Cyclosporine | Tacrolimus
Started | 10 | 25
Completed | 10 | 23
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporine | Tacrolimus | Total
Number analyzed (Participants) | 10 | 25 | 35
Age, Continuous [Median (Full Range); unit: years] | 64.5 [52 to 69] | 61 [27 to 69] | 62 [27 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 6 | 16 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 1 | 6 | 7
  Spain | 3 | 9 | 12
  Poland | 0 | 7 | 7
  Italy | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After the End of Treatment (SVR 12)
Description: Participants were considered to have achieved SVR12 if hepatitis C virus ribonucleic acid (HCV RNA) levels were less than (<) 25 international unit per milliliter (IU/mL) detectable or undetectable at 12 weeks after the end of treatment.
Time Frame: Week 36
Population: Intent to treat (ITT) analysis set included all enrolled participants who took at least 1 dose of investigational medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Tacrolimus
Number analyzed (Participants) | 10 | 25
percentage of participants | 100 [69.2 to 100] | 88 [68.8 to 97.5]

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 Weeks After the End of Treatment (SVR 4)
Description: Participants were considered to have achieved SVR4 if HCV RNA levels were (<) 25 IU/mL detectable or undetectable at 4 weeks after the end of treatment.
Time Frame: Week 28
Population: ITT analysis set included all enrolled participants who took at least 1 dose of investigational medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Tacrolimus
Number analyzed (Participants) | 10 | 25
percentage of participants | 100 [69.2 to 100] | 88 [68.8 to 97.5]

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks After the End of Treatment (SVR 24)
Description: Participants were considered to have achieved SVR 24 if hepatitis C virus ribonucleic acid (HCV RNA) levels were (<) 25 IU/mL detectable or undetectable at 24 weeks after the end of treatment.
Time Frame: Week 48
Population: ITT analysis set included all enrolled participants who took at least 1 dose of investigational medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Tacrolimus
Number analyzed (Participants) | 10 | 25
percentage of participants | 100 [69.2 to 100] | 88 [68.8 to 97.5]

4. Secondary Outcome: Percentage of Participants With HCV RNA (< 25 IU/mL Undetectable) and HCV RNA < 25 IU/mL Detectable
Description: Percentage of participants with detectable and undetectable HCV RNA (<) 25 IU/mL during treatment at Weeks 2,4, 12, and 24 were reported.
Time Frame: Weeks 2, 4, 12, and 24
Population: ITT analysis set included all enrolled participants who took at least 1 dose of investigational medication.
Measure: Number; unit: percentage of participants
Arm/Group | Cyclosporine | Tacrolimus
Number analyzed (Participants) | 10 | 25
percentage of participants
  Week 2: <25 IU/mL detectable | 30 | 36
  Week 2: <25 IU/mL undetectable | 10 | 12
  Week 4: <25 IU/mL detectable | 30 | 24
  Week 4: <25 IU/mL undetectable | 70 | 68
  Week 12: <25 IU/mL detectable | 0 | 0
  Week 12: <25 IU/mL undetectable | 100 | 96
  Week 24: <25 IU/mL detectable | 0 | 0
  Week 24: <25 IU/mL undetectable | 100 | 100

5. Secondary Outcome: Percentage of Participants With HCV RNA (<) 100 IU/mL at Week 4
Description: Percentage of participants with HCV RNA (<) 100 IU/mL at week 4 were reported.
Time Frame: Week 4
Population: ITT analysis set included all enrolled participants who took at least 1 dose of investigational medication.
Measure: Number; unit: percentage of participants
Arm/Group | Cyclosporine | Tacrolimus
Number analyzed (Participants) | 10 | 25
percentage of participants | 100 | 100

6. Secondary Outcome: Number of Participants With On-Treatment Failure
Description: On-treatment failure is defined as participants who did not achieve SVR12 and with confirmed detectable HCV RNA at the actual end of treatment. This was to include participants with: 1) Viral breakthrough, defined as a confirmed increase of greater than (>)1 log10 in HCV RNA from nadir, or confirmed HCV RNA of >100 IU/mL in participants whose HCV RNA had previously been <lower limit of quantification (LLOQ) while on treatment; 2) Other with confirmed detectable HCV RNA at the actual end of treatment (example, completed, discontinued due to adverse events (AEs), withdrawal of consent).
Time Frame: Up to Week 24 after actual EOT (week 24)
Population: ITT analysis set included all enrolled participants who took at least 1 dose of investigational medication.
Measure: Number; unit: participants
Arm/Group | Cyclosporine | Tacrolimus
Number analyzed (Participants) | 10 | 25
participants | 0 | 3

7. Secondary Outcome: Number of Participants With Viral Breakthrough
Description: Viral breakthrough is defined as a confirmed increase of >1 log10 IU/mL in HCV RNA level from the lowest level reached, or a confirmed HCV RNA level of >100 IU/mL in participants whose HCV RNA levels had previously been below the limit of quantification (<25 IU/mL detectable) or undetectable (<25 IU/mL undetectable) while on study treatment.
Time Frame: Up to week 24
Population: ITT analysis set included all enrolled participants who took at least 1 dose of investigational medication.
Measure: Number; unit: participants
Arm/Group | Cyclosporine | Tacrolimus
Number analyzed (Participants) | 10 | 25
participants | 0 | 3

8. Secondary Outcome: Number of Participants With Viral Relapse
Description: Participants who did not achieve SVR12, with undetectable HCV RNA at the actual end of study drug treatment and confirmed HCV RNA greater than or equal to (>=) LLOQ during follow-up.
Time Frame: Up to Week 24 after actual EOT (week 24)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cyclosporine | Tacrolimus
Number analyzed (Participants) | 10 | 25
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 52 Weeks
Arm/Group | Cyclosporine | Tacrolimus
Serious Adverse Events (participants affected / at risk) | 4/10 | 4/25
Other Adverse Events (participants affected / at risk) | 10/10 | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine (N=10) | Tacrolimus (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 1 | 0
Genital Herpes (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic Encephalopathy (Nervous system disorders) | 0 | 1
Loss of Consciousness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Micturition Disorder (Renal and urinary disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine (N=10) | Tacrolimus (N=25)
Anaemia (Blood and lymphatic system disorders) | 7 | 11
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 3
Ocular Icterus (Eye disorders) | 1 | 1
Visual Acuity Reduced (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Aphthous Stomatitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Lip Dry (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3
Tongue Dry (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Asthenia (General disorders) | 5 | 7
Fatigue (General disorders) | 2 | 1
Gait Disturbance (General disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 2
Mucous Membrane Disorder (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 2
Oral Candidiasis (Infections and infestations) | 0 | 2
Oral Herpes (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 4
Restless Legs Syndrome (Nervous system disorders) | 1 | 0
Anger (Psychiatric disorders) | 1 | 1
Hallucination, Visual (Psychiatric disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Vulvovaginal Pain (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.